CLINICAL TRIAL: NCT03193346
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled Study to Evaluate the Efficacy and Safety of BOTOX® (Botulinum Toxin Type A) as Headache Prophylaxis in Chinese Patients With Chronic Migraine
Brief Title: BOTOX® (Botulinum Toxin Type A) as Headache Prophylaxis in Chinese Participants With Chronic Migraine
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Corporation Decision
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1313-301-008
Record Dates: First submitted 2017-06-19; First posted 2017-06-20 (Actual); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Migraine Disorders
MeSH Terms: conditions — Migraine Disorders | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BOTOX® (Experimental): BOTOX® (botulinum toxin Type A) 155U to 195U intramuscular (IM) injections in head/neck areas at Day 0 and Week 12.
  Interventions: Biological: botulinum toxin Type A
- Placebo (Placebo Comparator): Placebo matching BOTOX® [Sodium chloride 0.9 milligrams (mg)] IM injections in head/neck areas at Day 0 and Week 12.
  Interventions: Drug: placebo (sodium chloride 0.9 mg)

INTERVENTIONS:
Biological: botulinum toxin Type A — Botulinum toxin Type A (BOTOX®) 155U to 195U IM injections in head/neck areas.
  Other Names: BOTOX®; onabotulinumtoxinA
  Arms: BOTOX®
Drug: placebo (sodium chloride 0.9 mg) — Placebo matching BOTOX® [Sodium chloride 0.9 mg] IM injections in head/neck areas.
  Arms: Placebo

SUMMARY:
This study will evaluate the efficacy and safety of BOTOX® (Botulinum Toxin Type A) compared with placebo as headache prophylaxis in Chinese participants with chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic migraine prior to the baseline phase based on the revised criteria for chronic migraine listed in International Classification of Headache Disorders (ICHD)-3 beta (2013)
* Fifteen or more headache days during the 4-week baseline phase, with each day consisting of 4 or more hours of continuous headache
* Routine non-headache medications of stable dose and regimen for at least 1 month prior to the start of screening.

Exclusion Criteria:

* Participants diagnosed with any of the following headache disorders: Familial hemiplegic migraine, Sporadic hemiplegic migraine, Migraine with brainstem aura, Migrainous infarction, Chronic tension-type headache, Hypnic headache, Hemicrania continua, New daily-persistent headache and Recurrent painful ophthalmoplegic neuropathy
* Participants with a confirmed history of medication overuse headache
* Participants with a diagnosis of retinal migraine, persistent aura without infarction or migraine-triggered seizure
* Headache attributable to another disorder (eg, cervical dystonia, craniotomy, head/neck trauma)
* Use of any headache prophylactic medication within 28 days prior to the start of the screening
* Any medical condition that may put the patient at increased risk with exposure to Botulinum Toxin Type A, including diagnosed myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, or any other significant disease that might interfere with neuromuscular function
* Participants with a known or suspected Temporomandibular Disorder (TMD), including pain in or around the Temporomandibular Joint (TMJ)
* Participants with a concurrent diagnosis of fibromyalgia
* Previous treatment with botulinum toxin therapy for any reason, or immunization to any botulinum toxin serotype
* Acupuncture, transcutaneous electrical nerve stimulation (TENS), cranial traction, nociceptive trigeminal inhibition or occipital nerve block treatments, or injection of anesthetics or steroids into the study target muscles within 28 days prior to the start of the screening
* Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminaemia, esophageal or gastric varices or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-03 (Estimated); Primary Completion 2021-03-25 (Estimated); Study Completion 2021-03-25 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in the Frequency of Headache Days during 28-Day Period Ending with Week 24 | Baseline, Week 24
  Mean change from Baseline (28-days prior to first treatment) in frequency (number) of headache days during the 28-day period ending with Week 24. A headache day was defined as a calendar day [00:00 to 23:59] for which the participant reported ≥ 4 continuous hours of headache per patient diary.

SECONDARY OUTCOMES:
Change from Baseline in the Frequency of Headache Days during 28-Day Period | Baseline, Weeks 4, 8, 12, 16 and 20
  Mean change from Baseline (28-days prior to first treatment) in frequency (number) of headache days during the 28-day period ending with Weeks 4, 8, 12, 16 and 20. A headache day was defined as a calendar day [00:00 to 23:59] for which the participant reported ≥ 4 continuous hours of headache per patient diary.
Change from Baseline in the Frequency of Migraine/Probable Migraine Days during 28-Day Period | Baseline, Weeks 4, 8, 12, 16, 20 and 24.
  Mean change from Baseline (28-days prior to first treatment) in frequency (number) of migraine or probable migraine episodes during the 28-day period ending with Weeks 4, 8, 12, 16, 20 and 24. A Migraine or Probable Migraine day was defined as a calendar day [00:00 to 23:59] for which the patient reported ≥ 4 continuous hours of a migraine or probable migraine episode as per the patient diary.
Change from Baseline in the Number of Moderate/Severe Headache Days during 28-Day Period | Baseline, Weeks 4, 8, 12, 16, 20 and 24
  Mean change from Baseline (28-days prior to first treatment) in frequency (number) of headache days during the 28 day period ending with Weeks 4, 8, 12, 16, 20 and 24. A moderate/severe headache day is defined as a day (00:00 to 23:59) when a participant reported 4 or more continuous hours of headache and reported a maximum severity of moderate or severe per patient diary among all headache episodes that occurred on that day.
Change from Baseline in Total Cumulative Hours of Headache Days during 28-Day Period | Baseline, Weeks 4, 8, 12, 16, 20 and 24
  Mean change from Baseline (28-days prior to first treatment) in the total cumulative hours of headache days during the 28-day period ending with Weeks 4, 8, 12, 16, 20 and 24. A headache day is defined as a day (00:00 to 23:59) with 4 or more continuous hours of headache per patient diary.

CONTACTS AND LOCATIONS:
Overall Officials: Arlene Lum, Study Director — Allergan

REFERENCES:
- See also: More Information — http://allerganclinicaltrials.com